CLINICAL TRIAL: NCT03320447
Title: Long-term Efficacy of Ablative Fractional Laser-assisted Photodynamic Therapy for Treatment of Lower Extremity Bowen's Disease: A Prospective, Randomized, Controlled Trial With 5-year Follow up
Brief Title: Long-term Efficacy of Ablative Fractional Laser-assisted Photodynamic Therapy for Treatment of Lower Extremity Bowen's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Song Ki-Hoon, Associate professor, Dong-A University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: DAUderma-09
Record Dates: First submitted 2017-10-19; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Bowen's Disease
Keywords: ablative fractional laser; photodynamic therapy; protoporphyrin IX; methy-aminolevulinate
MeSH Terms: conditions — Bowen's Disease | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAL-PDT (Experimental): Patients were randomly assigned to receive either AFL-PDT or MAL-PDT in a 1:1 ratio. As result, the patients were randomized to treatment with AFL-PDT or MAL-PDT
  Interventions: Drug: methyl-aminolevulinate application; Device: Illuminating using red light-emitting diode lamps
- AFL-PDT (Experimental): Patients were randomly assigned to receive either AFL-PDT or MAL-PDT in a 1:1 ratio. As result, the patients were randomized to treatment with AFL-PDT or MAL-PDT
  Interventions: Drug: lidocaine-prilocaine 5% cream application; Device: 2940-nm Er:YAG AFL pretreatment; Drug: methyl-aminolevulinate application; Device: Illuminating using red light-emitting diode lamps

INTERVENTIONS:
Drug: lidocaine-prilocaine 5% cream application — The lesions were then cleansed with saline gauze, and a lidocaine-prilocaine 5% cream (EMLA®; Astra Pharmaceuticals, LP, Westborough, MA, USA) was applied to the treatment area for 30 min under occlusion
  Arms: AFL-PDT
Device: 2940-nm Er:YAG AFL pretreatment — After the anesthetic cream was removed, AFL was performed using a 2940-nm Er:YAG AFL (Joule; Sciton, Inc., Palo Alto, CA, USA) with a 500 µm ablation depth, level 1 coagulation, 22% treatment density, and a single pulse
  Arms: AFL-PDT
Drug: methyl-aminolevulinate application — Immediately after the AFL, a 1-mm thick layer of methyl-aminolevulinate (16% Metvix® cream; PhotoCure ASA, Oslo, Norway) was applied to the lesion and to 5 mm of the surrounding healthy tissue. The area was covered with an occlusive dressing (Tegaderm; 3M, Co., Saint Paul, MN, USA) for 3 h, after which the remaining cream was removed with saline gauze, and the red fluorescence of porphyrins was visualized with Wood's light.
Device: Illuminating using red light-emitting diode lamps — Each treatment area was then separately illuminated using red light-emitting diode lamps (Aktilite CL128; Galderma S.A., Bruchsal, Germany) with peak emission at 632 nm and a total light dose of 37 J/cm2. Areas scheduled to receive MAL-PDT received the second treatment 7 days later. During the illumination, patients were asked to evaluate pain intensity using an 11-point visual analog scale.

SUMMARY:
Er:YAG ablative fractional laser-assisted methyl aminolevulinate photodynamic therapy (AFL-PDT) has shown significantly higher efficacy and a lower recurrence rate at 12 months than methyl aminolevulinate photodynamic therapy (MAL-PDT) for treatment of Bowen's disease (BD). However, long-term follow up data are not available.

DETAILED DESCRIPTION:
To compare the long-term efficacy and recurrence rates of AFL-PDT and standard MAL-PDT for the treatment of lower extremity BD.

ELIGIBILITY:
Inclusion Criteria:

* •Patients aged 18 years or more who diagnosed as bowen's disease

Exclusion Criteria:

* pregnancy or lactation
* active systemic infectious disease
* other inflammatory, infectious, or neoplastic skin diseases in the treated area
* allergy to MAL,other topical photosensitizers, or excipients of the cream
* history of photosensitivity
* use of immunosuppressive or photosensitizing drugs
* participation in any other investigational study in the preceding 30 days
* history or indicators of poor compliance
* Histological findings of acantholysis, desmoplasia, perineural or lymphovascular invasion, and echographic features of regional lymph node metastasis were the disease-specific exclusion criteria

Ages: 42 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10-30 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Difference of short-term complete response (CR) rate between AFL-PDT and MAL-PDT | Short-term CR rate was evaluated at 3 months
  The response was classified as either complete response (complete disappearance of the lesion) or incomplete response (incomplete disappearance of the lesion)
Difference of long-term complete response (CR) rate between AFL-PDT and MAL-PDT | Long-term CR rate was evaluated at 60 months
  The response was classified as either complete response (complete disappearance of the lesion) or incomplete response (incomplete disappearance of the lesion)
Difference of long-term recurrence rate between AFL-PDT and MAL-PDT at 60 months | Recurrent rate was evaluated at 60 months
  In all cases of complete response, the patients were reviewed at 60 months to check for recurrence. Post-therapy punch biopsies were performed when there was doubt concerning incomplete-response and clinical recurrence

SECONDARY OUTCOMES:
Difference of the cosmetic outcome between AFL-PDT and MAL-PDT | Cosmetic outcome was assessed by each investigator for all lesions that achieved a complete response at 60 months
  The overall cosmetic outcome was assessed by each investigator for all lesions that achieved complete response at 60 months, and was graded using a 4-point scale: excellent (only slight occurrence of redness or change in pigmentation), good (moderate redness or change in pigmentation), fair (slight to moderate scarring, atrophy, or induration), or poor (extensive scarring, atrophy, or induration)

OTHER OUTCOMES:
Differences of Adverse events(erythema, burning sensation, swelling, bleeding) between AFL-PDT and MAL-PDT | Within 60 months after each treatment
  Adverse events reported by the patients were noted at each follow-up visit, including severity, duration, and need for additional therapy. All events due to PDT were described as phototoxic reactions(e.g erythema, burning sensation, swelling, bleeding)

IPD SHARING:
Plan to Share IPD: No